CLINICAL TRIAL: NCT00941005
Title: The Effect of Electroacustimulation on Postoperative Nausea, Vomiting and Pain in Outpatient Plastic Surgery Patients: A Prospective, Randomized, Blinded Clinical Trial
Brief Title: The Effect of Electroacustimulation on Postoperative Nausea, Vomiting and Pain in Outpatient Plastic Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-2007-0100
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electroacustimulation (Experimental): Received electroacustimulation at the wrist using a small, battery-powered electroacustimulation device.
  Interventions: Device: Electroacustimulation
- Control (Sham Comparator): Received a device that was not turned on.
  Interventions: Device: Electroacustimulation

INTERVENTIONS:
Device: Electroacustimulation — Electroacustimulation (EAS) is a derivative form of acupuncture therapy where a small current of electricity instead of a needle is used to stimulate an acupoint on the human body in an effort to create therapeutic effects.
  Other Names: ReliefBand (Aeromedix, Jackson, WY)

SUMMARY:
Introduction: Current rates of postoperative nausea and vomiting (PONV) experienced by outpatient surgery patients are as high as 20-30%. Electroacustimulation (EAS) therapy has been demonstrated to be effective in controlling these symptoms, but trials identifying their efficacy in the outpatient surgery population are lacking. This study integrates conventional pharmacotherapy with alternative medicine in prevention of PONV.

Materials and Methods: One hundred twenty two patients undergoing surgery procedures at an outpatient surgery center were randomized to two treatment arms. The first arm was standardized pharmacologic PONV prevention typical for patients undergoing outpatient surgery, while the second arm employed the use of ReliefBand, an FDA-approved electroacustimulation (EAS) device with pharmacologic treatment to relieve symptoms of PONV and pain. EAS is a derivative of acupuncture therapy that uses a small electrical current to stimulate acupuncture points on the human body and is thought to relieve nausea, vomiting and pain. Outcomes measured were post-op questionnaires evaluating pain and nausea symptoms, emetic events, the need for rescue medications and the time to discharge.

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery at the University of Wisconsin outpatient surgery center

Exclusion Criteria:

* pregnancy
* currently experiencing menstrual symptoms
* cardiac pacemaker
* previous experience with acupuncture therapy
* pharmacologic treatment for nausea or vomiting in the 24 hours prior to surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karol A Gutowski, MD, Principal Investigator — Endeavor Health
Locations (1):
- Transformations Surgery Center, Middleton, Wisconsin, United States

REFERENCES:
- [Background] Gan TJ, Jiao KR, Zenn M, Georgiade G. A randomized controlled comparison of electro-acupoint stimulation or ondansetron versus placebo for the prevention of postoperative nausea and vomiting. Anesth Analg. 2004 Oct;99(4):1070-1075. doi: 10.1213/01.ANE.0000130355.91214.9E. PMID 15385352
- [Result] Larson JD, Gutowski KA, Marcus BC, Rao VK, Avery PG, Stacey DH, Yang RZ. The effect of electroacustimulation on postoperative nausea, vomiting, and pain in outpatient plastic surgery patients: a prospective, randomized, blinded, clinical trial. Plast Reconstr Surg. 2010 Mar;125(3):989-94. doi: 10.1097/PRS.0b013e3181ccdc23. PMID 20195124

RESULTS

PARTICIPANT FLOW:
Groups:
- Electroacustimulation: Received electroacustimulation at the wrist using a small, battery-powered electroacustimulation device, ReliefBand as well as pharmacologic measures.
  Electroacustimulation: Electroacustimulation (EAS) is a derivative form of acupuncture therapy where a small current of electricity instead of a needle is used to stimulate an acupoint on the human body in an effort to create therapeutic effects.
- Control: Sham electroacustimulation device (turned off)
  Standardized pharmacologic postoperative nausea and vomiting prevention typical for patients undergoing outpatient surgery
Period: Overall Study
Arm/Group | Electroacustimulation | Control
Started | 61 | 61
Completed | 61 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Raw data no longer exist for this study. We have done our due diligence to populate this record with data provided in the publication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Electroacustimulation | Control | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Customized [Number; unit: participants]
  Data no longer exists | NA — data no longer exists | NA — data no longer exists | NA — data no longer exists
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data no longer exist for this study | NA — Data no longer exist for this study | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data no longer exist for this study | NA — Data no longer exist for this study | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 61 | 61 | 122

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Nausea Scores
Description: Nausea is scored on a scale of 1-10 where 1 is least nauseated and 10 is severely nauseated. Nausea scores will be collected 30, 60, and 120 minutes after surgery.
Time Frame: 24 hours
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Electroacustimulation | Control
Number analyzed (Participants) | 61 | 61
participants
  30 min post-op | NA — Data cannot be confirmed | NA — Data cannot be confirmed
  60 min post-op | NA — Data cannot be confirmed | NA — Data cannot be confirmed
  120 min post-op | NA — Data cannot be confirmed | NA — Data cannot be confirmed

2. Primary Outcome: Incidence of Post-operative Emetic Events
Time Frame: 24 hours
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: incidence of emetic events
Arm/Group | Electroacustimulation | Control
Number analyzed (Participants) | 61 | 61
incidence of emetic events | 0 (0) | 0 (0)

3. Primary Outcome: Number of Participants With Post-operative Need for Rescue Medications
Time Frame: 24 hours
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacustimulation | Control
Number analyzed (Participants) | 61 | 61
Participants | NA — Data cannot be confirmed | NA — Data cannot be confirmed

4. Primary Outcome: Time to Participant Discharge
Time Frame: 24 hours
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Electroacustimulation | Control
Number analyzed (Participants) | 61 | 61
minutes | NA (NA) — Data cannot be confirmed | NA (NA) — Data cannot be confirmed

5. Primary Outcome: Phone Survey of Nausea / Vomiting Symptoms 24 Hours Post-op
Description: Phone survey of nausea/vomiting symptoms was administered on postoperative day 1. The survey consists of 8 questions, including: 1) a query about whether or not participant has experienced nausea since returning home; 2) rate nausea severity on a scale of 1-10 (where 10 is the most severe); 3) a query about satisfaction of nausea control; 4) a question asking if they would use the same post-op nausea treatment again; 5) a query about what activities the participant has been unable to do since surgery; 6) whether or not the participant has taken prescription medicine for treatment of nausea since returning home; 7) whether or not participant has taken prescription medicine for treatment of pain since returning home; and 8) if yes for 6-7, which medications.
Time Frame: 24 hours post-op
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Electroacustimulation | Control
Number analyzed (Participants) | 61 | 61
score on a scale | NA (NA) — Data cannot be confirmed | NA (NA) — Data cannot be confirmed

6. Secondary Outcome: Postoperative Pain Scores
Description: Participants will evaluate their postoperative pain score on a scale of 1-10 where 1 is the least pain and 10 is the most severe pain. Pain scores will be evaluated at 30, 60, and 120 minutes postop.
Time Frame: 24 hours
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Electroacustimulation | Control
Number analyzed (Participants) | 61 | 61
score on a scale
  30 min post-op | NA (NA) — Data cannot be confirmed | NA (NA) — Data cannot be confirmed
  60 min post-op | NA (NA) — Data cannot be confirmed | NA (NA) — Data cannot be confirmed
  120 min post-op | NA (NA) — Data cannot be confirmed | NA (NA) — Data cannot be confirmed

7. Secondary Outcome: Number of Participants Who Took Pain Medicine in the First 24 Hours Post-op
Description: Phone survey of post-op pain medication usage was administered on postoperative day 1.
Time Frame: 24 hours post-op
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Electroacustimulation | Control
Number analyzed (Participants) | 61 | 61
Participants | NA — Data cannot be confirmed | NA — Data cannot be confirmed

ADVERSE EVENTS:
Time Frame: up to 24 hours post-operatively
Description: Raw data no longer exist for this study. We have done our due diligence to populate this record with data provided in the publication. There is no evidence that Adverse Events Data was monitored.
Arm/Group | Electroacustimulation | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Raw data from which to report summary results no longer exist for this study. Outcomes were published and the data were represented in graphs. We have done our due diligence to populate this record with data provided in the publication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes